CLINICAL TRIAL: NCT00493558
Title: A Consecutive Case Series of One-Level Lumbar Fusions With Pedicle Screw Instrumentation and the Trabecular Metal™ Intervertebral Cage Using Roentgen Stereophotogrammetric Analysis (RSA)
Brief Title: Spine Research With Roentgen Stereophotogrammetric Analysis
Acronym: SpineRSA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Principal Investigator, William Oxner, Principal Investigator, Nova Scotia Health Authority
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDHA018
Record Dates: First submitted 2007-06-27; First posted 2007-06-28 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Spondylolisthesis; Degenerative Lumbar Disc Disease; Spinal Stenosis
Keywords: Roentgen Stereophotogrammetric Analysis; Trabecular Metal Posterior Lumbar Interbody Cage; Posterior Lumbar Interbody Fusion Cage; Posterior Lumbar spine fusion surgery
MeSH Terms: conditions — Spondylolisthesis; Spinal Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Trabecular Metal Intervertebral Cage with RSA beads — Roentgen Stereophotogrammetric Analysis beads will be inserted at time of implant of the Trabecular Metal Intervertebral Cage.

SUMMARY:
The purpose of this study is to gather information on the effectiveness of a new spine implant for patients who require spinal fusion surgery. Based on this information, we hope to create a standard of good performance, or benchmark, against which future studies on this spine implant can be compared. By creating this benchmark we hope to improve care for patients who require spinal fusion surgery.

DETAILED DESCRIPTION:
For patients in whom a spinal fusion is indicated, the posterior lumbar interbody fusion (PLIF) may be recommended to restore stability to the affected spinal segment1. Pioneered by a Dr.Cloward in the 1940s to treat painful intervertebral discs damaged by degeneration, PLIF involves removal of the entire nuclear portion of the disc and subsequent replacement with multiple blocks of transplanted bone. The purpose of the fusion is to eliminate or reduce the amount of the motion at the affected site, and, therefore, the source of pain.

Four major intervertebral cages have been approved by the Food and Drug Administration (FDA) for use in humans: the Brantigan Interbody fusion Cage, the Ray Threaded Fusion Cage, the Bagby and Kuslich cage, and, most recently, the Trabecular Metal™ Cage. Comprised of 98 percent tantalum and 2 percent vitreous carbon, Trabecular Metal™ has the highest coefficient of friction of any implant material on the market, allowing for optimal initial implant-bone fit. Furthermore, the unique porous structure of Trabecular Metal™ provides significantly more space for tissue ingrowth to occur, facilitating a more cohesive implant-bone interface as well as long-term stability of the implant.

Long-term follow up data on the efficacy of the Brantigan Interbody fusion cage, Ray Threaded Fusion cage, and Bagby and Kuslich cages are limited, with the most rigorous studies (i.e. controlled prospective studies) typically providing outcomes approximately 2 years post-surgery. Overall, these studies show that, while existing intervertebral cages have made significant advances in terms of addressing the disadvantages associated with traditional bone grafting/fixation techniques, problems continue to persist. Through comprehensive and accurate clinical evaluation of the Trabecular Metal™ intervertebral cage, the Research Team hopes to document advances in the PLIF technique, thereby informing current research as well as clinical practice.

The primary goal of the proposed research is to gather data on the clinical efficacy of the Trabecular Metal™ Posterior Lumbar Interbody Fusion (PLIF) cage with pedicle screw instrumentation for the treatment of one-level lumbar spine fusions. Based on this pilot data, we hope to establish a level of acceptable clinical performance for the Trabecular Metal™ cage, a benchmark against which subsequent investigations can be compared.

Direct surgical exploration is considered the most reliable method for accurately determining fusion success, both from a structural and functional perspective, following spinal fusion surgery. Unfortunately, this method is highly invasive, costly and seldom used. Furthermore, surgical exploration does not provide any longitudinal information as to the stability of the implant, including the monitoring of any occurrence of migration.

In contrast, Roentgen Stereophotogrammetric Analysis(RSA)can detect the presence or absence of mobility between intervertebral segments (i.e. functional stability of the fusion) with a high degree of accuracy. RSA is a radiographic technique that uses small tantalum balls implanted into the patient's bone to measure micromotion (<1 mm) at the bone - implant interface, something which is not possible to do reliably using regular x-ray techniques. RSA provides a method for detecting inferior implant designs or cement formulations using only a small number of patients before release of these products into large clinical trials.

RSA has been in use for several decades,and its safety is well documented.A computerized, digital RSA system has recently been installed and calibrated at our center. Its measurement capabilities have been rigorously validated, and it is currently being used to assess a new knee implant design. Expansion of the system to include spine RSA can be easily accomplished.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 20 years of age
* Clinical and radiologic history of spondylolisthesis (no greater than grade 1)
* Spinal stenosis for which conservative treatment has failed
* Degenerative disc disease, characterized by one or more of the following:

  * instability (defined as angular motion > 5° and/or translation > 4mm, based on Flex/Ext radiographs)
  * osteophyte formation
  * decreased disc height
  * thickening of ligamentous tissue
  * disc degeneration or herniation
  * facet joint degeneration

Exclusion Criteria:

* Fusion at more than one level
* Non-fusion surgery at the involved level
* Previously diagnosed with osteopenia, osteoporosis, or osteomalacia to a degree that spinal instrumentation would be contraindicated
* Patients with a highly-communicable disease, inflammatory or auto-immune based joint disease
* Those with a history of endocrine or metabolic disorders known to affect osteogenesis (e.g. Paget's disease, renal osteodystrophy, Ehlers-Danios syndrome or osteogenesis imperfecta)
* Patients with a documented titanium or tantalum alloy allergy or intolerance
* Patients currently receiving active treatment for cancer or treatment with steroids such as cortisone
* Patients with significant medical history that, in the Investigator's opinion, would not make them a good study candidate

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Spinal fusion and the rate of fusion and maintenance of spinal alignment will be assessed | 6 weeks, 3, 6, 12, and 24months.

SECONDARY OUTCOMES:
Subjective outcome questionnaires will be used to characterize the patient sample used for the study to allow for comparisons to other treatments for this condition in the future. | 3, 6, 12, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Wm Oxner, M.D., Principal Investigator — Capital District Health Authority, QEII Health Science Centre, & Dalhousie University, Halifax. Nova Scotia,Canada
Locations (1):
- Capital District Health Authority, QEII Health Sciences Centre,& Dalhousie University, Halifax, Nova Scotia, Canada